CLINICAL TRIAL: NCT06169956
Title: Neoadjuvant Nivolumab (OPDIVO®) in Combination With Platinum-Based Chemotherapy for Non-Metastatic NSCLC: A German, Nationwide, Prospective, Observational, Multicenter Study in Patients Scheduled to Receive 3 Cycles Nivolumab in Combination With Platinum-Based Chemotherapy for Non-Metastatic (Stage and PD-L1 Expression According to Label) Non-Small Cell Lung Cancer
Brief Title: An Observational Study to Evaluate Neoadjuvant Nivolumab (OPDIVO®) in Combination With Platinum-Based Chemotherapy in Non-Metastatic Non-Small Cell Lung Cancer Participants in Germany
Acronym: NENI
Status: Recruiting | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-1210
Record Dates: First submitted 2023-11-17; First posted 2023-12-14 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Resectable Non-small Cell Lung Cancer
MeSH Terms: interventions — Platinum Compounds

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants receiving neoadjuvant nivolumab in combination with platinum-based chemotherapy
  Interventions: Drug: Neoadjuvant nivolumab in combination with platinum-based chemotherapy

INTERVENTIONS:
Drug: Neoadjuvant nivolumab in combination with platinum-based chemotherapy — Neoadjuvant treatment of resectable non-small cell lung cancer with nivolumab in combination with chemotherapy according to current summary of product characteristics

SUMMARY:
The purpose of this observational study is to collect and evaluate real-world data to assess the effectiveness of neoadjuvant nivolumab when given in combination with platinum-based chemotherapy in participants with early-stage, resectable non-small cell lung cancer (NSCLC) in Germany

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Diagnosis of non-metastatic non-small cell lung cancer with tumor Programmed death-ligand 1 (PD-L1) expression level of 1% or more (tumor proportion score (TPS); according to label approved in the European Union)
* Decision to initiate a neoadjuvant treatment with nivolumab plus platinum-based chemotherapy for treatment of non-small cell lung cancer according to current Summary of product characteristics and independent of the study
* Willing to complete patient-reported outcome questionnaires and sufficient understanding of the German language
* Signed written informed consent
* Other criteria according to current Summary of product characteristics

Exclusion Criteria:

* Current primary diagnosis of cancer other than non-small cell lung cancer that requires systemic or other treatment
* Other contraindications according to current Summary of product characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants aged ≥ 18 years of age or older who are diagnosed with resectable non-small cell lung cancer at high risk of recurrence and whose tumors have programmed death-ligand 1 (PD-L1) expression ≥ 1%
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-11-30 (Actual); Primary Completion 2030-09-30 (Estimated); Study Completion 2030-09-30 (Estimated)

PRIMARY OUTCOMES:
Event-free survival | Up to 5 years

SECONDARY OUTCOMES:
Pathologic complete response (pCR) rate | Up to 5 years
Rate of major pathologic response (MPR) | Up to 5 years
Rate of partial pathologic response (pPR) | Up to 5 years
Rate of pathologic non-responder | Up to 5 years
Rate of tumor response | Up to 5 years
  Classified as complete response (CR), partial response (PR), stable disease (SD), progressive disease (PD)
Participant age | Baseline
Participant sex | Baseline
Participant insurance status | Baseline
Participant employment status | Baseline
Participant height in cm | Baseline
Participant weight in kg | Baseline
Eastern Cooperative Oncology Group Performance Status (ECOG-PS) | Baseline and up to 5 years
  ECOG-PS score of 0 = Fully active, able to carry on all pre-disease performance without restriction. ECOG-PS score of 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work. ECOPG-PS score of 2 = Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours. ECOG-PS score of 3 = Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours. ECOG-PS score of 4 = Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair. ECOG-PS score of 5 = Dead
Participant medical history | Baseline
Participant history of smoking | Baseline
Participant concomitant treatments | Baseline and during neoadjuvant nivolumab plus platinum-based chemotherapy, up to 5 years
Participant subsequent treatments | Up to 5 years
Date of initial diagnosis of NSCLC | Baseline
Primary tumor assessed by histology subtype | Baseline
Tumor stage assessed by tumor node metastasis (TNM; stage IB-IIIA) | Baseline
Location of primary tumor | Baseline
Date of local relapse | Baseline to end of study, up to 5 years
Location of metastases | Baseline to end of study, up to 5 years
Date of metastatic diagnosis | Baseline to end of study, up to 5 years
Tumor size assessed by medical imaging using x-rays, computed tomography (CT), magnetic resonance imaging (MRI), ultrasound, bone scintigraphy, positron emission tomography-computed tomography (PET- CT) | Up to 5 years
Tumor location assessed by medical imaging using x-rays, computed tomography (CT), magnetic resonance imaging (MRI), ultrasound, bone scintigraphy, positron emission tomography-computed tomography (PET- CT) | Up to 5 years
Number of participants with abnormal hematology results | Up to 5 years
Number of participants with abnormal clinical chemistry results | Up to 5 years
Number of participants with abnormal biomarker results | Baseline to end of study, up to 5 years
Type of surgery | Up to 5 years
Completeness of resection assessed by residual tumor classification | Up to 5 years
  R0: no residual tumor, R1: microscopic residual tumor, R2: macroscopic residual tumor, Rx: unknown
Number of participants with tumor resection | Up to 5 years
Extend of resection (R0/R1/R2) | Up to 5 years
Number of lymph nodes resected | Up to 5 years
Surgical approach | Up to 5 years
  Thoracotomy, minimal invasive (video-assisted thoracoscopic surgery [VATS], robotic-assisted thoracic surgery [RATS]), minimal invasive to thoracotomy (conversion)
Length of hospital stay following surgery | From surgery to discharge from hospital, assessed up to 5 years
Incidence of adverse events | Up to 5 years
Severity of adverse events graded by Common Terminology Criteria for Adverse Events (CTCAE) V5.0 | Up to 5 years
Patient-reported health-related Quality of Life assessed by using the validated European Quality of Life 5 Dimension 3 Level (EQ-5D-3L) questionnaire | Up to 5 years
  EQ-5D-3L summary index: 1 represents perfect health, 0 represents death, negative values represent health states considered worse than death
Time to next treatment | Up to 5 years
  Time between end of primary treatment (neoadjuvant treatment + surgery + if needed by physician's assessment adjuvant therapy) to start of next treatment)
Dosing of nivolumab | Up to 5 years
Treatment regimens | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Klinikverbund Allgaeu, Kempten (Allgäu), Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/safety/recalls-market-withdrawals-safety-alerts